CLINICAL TRIAL: NCT01289431
Title: Dose Ranging Study to Evaluate the Safety and Efficacy of Mapracorat Ophthalmic Formulation, in Subjects With Allergic Conjunctivitis Compared to Vehicle in a Conjunctival Allergen Challenge (CAC).
Brief Title: Mapracorat Ophthalmic Formulation in Subjects With Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 685
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mapracorat (Experimental)
  Interventions: Drug: Mapracorat
- Mapracorat Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Mapracorat — administered daily to each eye for 2 weeks following allergen challenge using a CAC model
  Arms: Mapracorat
Drug: Vehicle — administered daily to each eye for 2 weeks following allergen challenge using a CAC model
  Arms: Mapracorat Vehicle

SUMMARY:
The objective of this study is to evaluate the dose response, and efficacy of Mapracorat ophthalmic formulation compared to its vehicle for the prevention of symptoms and signs associated with allergic conjunctivitis using a conjunctival allergen challenge (CAC) model.

ELIGIBILITY:
Inclusion Criteria:

* positive history of ocular allergies and a positive skin test reaction
* positive bilateral CAC reaction

Exclusion Criteria:

* have known contraindications or sensitivities to the use of any of the study medications(s) or their components.
* have any ocular condition or significant illness that, in the opinion of the investigator, could affect the subject's safety or trial parameters.
* had ocular surgical intervention within three (3) months prior to Visit 1 or during the study and/or a history of refractive surgery within the past 3 months;
* a known history of retinal detachment, diabetic retinopathy, or active retinal disease;
* the presence of an active ocular infection or positive history of an ocular herpetic infection at any visit.
* use of any disallowed medications during the period indicated prior to Visit 1 and during the study.
* have planned surgery during the trial period or within 30 days after.
* have an intraocular pressure that is less than 5 mmHg or greater than 22 mmHg or any type of glaucoma at Visit 1

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ozden, OD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3% Once a Day; 2% Once a Day; 3% Once a Day; 0.3% Twice a Day; 2% Twice a Day; 3% Twice a Day: BOL-303242-X dosed in the eye
- Vehicle: Vehicle of BOL-303242-X dosed in the eye
Period: Overall Study
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle
Started | 34 | 34 | 34 | 33 | 34 | 33 | 34
Completed | 29 | 32 | 30 | 28 | 32 | 31 | 33
Not Completed | 5 | 2 | 4 | 5 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle | Total
Number analyzed (Participants) | 34 | 34 | 34 | 33 | 34 | 33 | 34 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (10.41) | 35.4 (13.62) | 37.7 (16.10) | 31.4 (11.46) | 36.0 (13.82) | 32.4 (12.03) | 35.1 (13.61) | 35.0 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 21 | 17 | 17 | 14 | 15 | 121
  Male | 16 | 15 | 13 | 16 | 17 | 19 | 19 | 115

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching was assessed by the participant on a 0-4 scale with half unit increments allowed. Lower scores indicate less ocular itching.
Time Frame: 8 hours
Population: Participants with results at the 8 hour timepoint are included, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle
Number analyzed (Participants) | 30 | 33 | 30 | 28 | 33 | 31 | 33
score on a scale | 1.71 (1.212) | 1.34 (0.757) | 2.11 (1.196) | 2.06 (0.880) | 1.65 (0.804) | 1.58 (0.842) | 2.28 (0.985)

2. Primary Outcome: Conjunctival Redness
Description: Conjunctival redness was assessed by the Investigator on a 0-4 scale with half unit increments allowed. Lower scores indicate less conjunctival redness.
Time Frame: 8 hours
Population: Participants with results at the 8 hour timepoint are included, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle
Number analyzed (Participants) | 30 | 33 | 30 | 28 | 33 | 31 | 33
score on a scale | 2.05 (0.757) | 1.56 (0.723) | 2.01 (0.791) | 1.82 (0.779) | 1.72 (0.828) | 1.81 (0.757) | 2.14 (0.631)

3. Secondary Outcome: Ciliary Redness
Description: The Investigator evaluated ciliary redness on a 0-4 scale with half unit increments allowed. A lower score is indicative of less ciliary redness.
Time Frame: 8 hours
Population: Participants with results at the 8 hour timepoint are included, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle
Number analyzed (Participants) | 30 | 33 | 30 | 28 | 33 | 31 | 33
score on a scale | 1.88 (0.903) | 1.39 (0.860) | 1.89 (0.875) | 1.60 (0.850) | 1.58 (0.915) | 1.65 (0.751) | 2.02 (0.780)

4. Secondary Outcome: Episcleral Redness
Description: Episcleral redness was evaluated by the Investigator using a 0-4 scale with half unit increments allowed. A lower score is indicative of less episcleral redness.
Time Frame: 8 hours
Population: Participants with results at the 8 hour timepoint are included, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle
Number analyzed (Participants) | 30 | 33 | 30 | 28 | 33 | 31 | 33
score on a scale | 2.11 (0.739) | 1.56 (0.735) | 2.07 (0.763) | 1.85 (0.805) | 1.79 (0.868) | 1.97 (0.772) | 2.25 (0.632)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | 0.3% Once a Day | 2% Once a Day | 3% Once a Day | 0.3% Twice a Day | 2% Twice a Day | 3% Twice a Day | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/33 | 0/34 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 1/34 | 0/34 | 4/34 | 1/33 | 2/34 | 2/33 | 7/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.3% Once a Day (N=34) | 2% Once a Day (N=34) | 3% Once a Day (N=34) | 0.3% Twice a Day (N=33) | 2% Twice a Day (N=34) | 3% Twice a Day (N=33) | Vehicle (N=34)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 2
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Instillation site abnormal sensation (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Instillation site pruritus (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.